# Practice Facilitation to Promote Evidence-based Screening and Management of Unhealthy Alcohol Use in Primary Care

# Research Participant Information and Consent Form

<u>Investigator & Sponsor</u>: Alex Kirst, MD, MPH (703) 389-2404, Agency for Healthcare Research and Quality

#### **Invitation to Participate**

You are invited to participate in a research on unhealthy alcohol use. This component of the study will include surveys on your clinic. This consent form is to assist you in deciding whether to participate in this study. This research is being conducted to learn more about how physicians communicate with patients regarding alcohol use and how to improve screening and interventions. If you agree to participate, you will be asked to complete two surveys and one exit interview. Both surveys and the interview will be completed verbally, in a group setting with your practice staff. One survey will be administered now and the second survey and exit interview will be administered at the end of the study in six months.

#### **Risks**

The main possible risk of participation is breach of confidentiality and privacy. The research team has implemented several procedures to minimize these risks.

## **Benefits**

This is a quality improvement study to help clinicians and practices how to better implement the US Preventive Services Task Force recommended preventive service of screening and counseling patients for unhealthy alcohol use. As a result of participating in this study, you and your office may do a better job of providing this recommended preventive services to your patients.

## **Costs and Payment**

There are no costs for participating in this study. There are no payments for participating in this research.

#### **Confidentiality**

The data in this study will be kept confidential. Your responses will be deidentified except for a code that will link survey results with your practice. The code, and your responses, will be held on a private, protected device. When analyzing your responses, researchers will not have access to the key code. No participant or practice names will be used when reporting information from survey results. The surveys responses will only be accessible to the researchers, and will be stored on a private, protected drive. Only aggregate results will be shared.

## **Voluntary Participation**

Participation in this study is voluntary at all times. Please ask the investigator or study staff to explain any information in this document that is not clear to you. You may choose not to participate or may revoke consent at any time. If you decide to withdraw, there will be no

penalty to you or your practice; data collected prior to withdrawal will be used for research, unless you request otherwise.

#### **Statement of Consent**

I have been provided with an opportunity to read this consent form carefully. All of the questions that I wish to raise concerning the study have been answered. I verbally agree to participate in this study.

For questions about this study, contact our office or Dr. Alex Krist or Dr. Alison Huffstetler, principal investigator and study lead, at (804) 827-2762; <a href="mailto:ahkrist@vcu.edu">ahkrist@vcu.edu</a>, or <a href="mailto:Alison.Huffstetler@vcuhealth.org">Alison.Huffstetler@vcuhealth.org</a>.

For questions about your rights as a research participant, or if you wish to discuss problems, concerns or questions, to obtain information, or to offer input about research, please contact the Office of Research Subjects Protection at Virginia Commonwealth University, PO Box 980568, Richmond, Virginia, 23298; (804) 827-2157;

https://research.vcu.edu/human research/volunteers.htm